CLINICAL TRIAL: NCT04349514
Title: A Natural History Study to TRACK Brain and Spinal Cord Changes in Individuals with Friedreich Ataxia (TRACK-FA)
Acronym: (TRACK-FA)
Status: Active, not recruiting | Type: Observational
Sponsor: Monash University (Other)
Collaborators: University of Minnesota (Other); RWTH Aachen University (Other); University of Campinas, Brazil (Other); Children's Hospital of Philadelphia (Other); University of Florida (Other); Friedreich's Ataxia Research Alliance (Other); McGill University (Other)
Responsible Party: Principal Investigator, Nellie Georgiou-Karistianis, Professor Nellie Georgiou-Karistianis, Monash University
Other Study IDs: TRACK-FA
Record Dates: First submitted 2020-04-01; First posted 2020-04-16 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-10

CONDITIONS: Friedreich Ataxia
Keywords: Neuroimaging; Longitudinal; Biomarkers; Natural history
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood sample (approximately 18-20ml) will be collected from each participant at the first assessment by a trained phlebotomist or clinician and processed immediately by research staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Friedreich ataxia: Individuals with a diagnosis of Friedreich ataxia.
  Interventions: Other: Natural history
- Control: Individuals without a diagnosis of Friedreich ataxia.
  Interventions: Other: Natural history

INTERVENTIONS:
Other: Natural history — Longitudinal observation of neuroimaging, clinical, and blood markers.

SUMMARY:
This is a natural history study prospectively investigating neuroimaging markers of disease progression in children and adults with Friedreich ataxia (FA). There will be three assessment periods (baseline, 12 and 24 months). The study will include approximately 200 individuals with FA and 100 matched controls recruited across the six international academic sites. Other assessments will include secondary clinical and cognitive markers, as well as exploratory blood markers.

DETAILED DESCRIPTION:
Friedreich ataxia (FA) is a multi-system progressive disorder with the most prevalent and prominent symptoms relating to dysfunction in the central and peripheral nervous system, including, loss of balance and coordination, frequent falls, loss of ambulation, dysarthria, dysphagia and loss of vision and hearing. Other symptoms include cardiomyopathy, diabetes, scoliosis and fatigue. Age of onset can vary but most often presents during childhood, ages 5-15 years.

There is currently no cure and no disease-modifying treatment. Drug candidates to potentially treat FA are under development; however, there is a lack of well- characterized neuroimaging biomarkers for testing their efficacy in clinical trials, hampering this process. Establishing disease-specific neuroimaging biomarkers to track disease progression requires high-quality longitudinal data from large cohorts of patients, compared to controls. In rare diseases, such as FA, this can only be achieved through multi-site collaboration.

The aim of TRACK-FA is to develop an FA neuroimaging dataset from brain and spinal cord that is suitable for assessing the potential value of neuroimaging biomarkers and providing a basis for instituting them in clinical trials. The dataset will comprise a range of neuroimaging measures to assess changes in spinal cord and brain regions that have previously shown to be compromised in individuals with FA. In addition to neuroimaging measures, TRACK-FA will also include clinical, cognitive data and biospecimen data. The TRACK-FA dataset will provide a unique opportunity for academic researchers in collaboration with industry partners to access the images, subsidiary data, and associated clinical data for community research.

This multi-centre study is a collaborative effort across six academic institutions, together with industry partners and the Friedreich's Ataxia Research Alliance USA (FARA).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 5 years
* Written informed consent provided
* Individuals with FA must have a genetic confirmation of diagnosis and be biallelic for a GAA repeat length > 55 in intron 1 of FXN and/or have a GAA repeat length > 55 in intron 1 of FXN in one allele and another type of mutation that is inferred to cause loss of function in the second FXN allele
* Individuals with FA must have an age of disease onset ≤ 25 years
* Individuals with FA must have a disease duration ≤ 25 years
* Individuals with FA must have a Friedreich Ataxia Rating Scale (FARS) Functional staging score of ≤ 5 and total modified FARS (mFARS) score of ≤ 65 on enrolment

Exclusion Criteria:

* Age < 5 years
* Unable to provide written informed consent
* Magnetic resonance contraindications (e.g. pacemaker or other metallic surgical implants)
* Presence of metallic dental braces
* Pregnancy (ascertained via a question or test as mandated at particular sites)
* Individuals with FA must not have acute or ongoing medical or other conditions that, after discussion between the Site Investigator and steering committee, is deemed to interfere with the conduct and assessments of the study
* Individuals with FA must not have another neurological condition apart from FA
* Individuals with FA must not have other neurologic conditions that, in the opinion of the Site Investigator, would interfere with the conduct and assessments of the study
* Controls must not have a diagnosed psychiatric or neurological condition
* Controls must not have acute or ongoing medical or other conditions that would interfere with the conduct and assessments of the study
* Controls must not be siblings of individuals with FA whose carrier status (i.e., confirmed carrier, confirmed non-carrier, or obligate carrier) is unknown.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of individuals aged 5 and above who either have a diagnosis of Friedreich ataxia (FA) or who do not (Controls). Controls will be healthy volunteers who are age- and gender-matched to the FA cohort.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Baseline dentate nuclei magnetic susceptibility | Baseline
  Magnetic susceptibility of the dentate nuclei will be measured using T2*-weighted multiecho magnetic resonance imaging and quantitative susceptibility mapping processing. Baseline dentate nuclei susceptibility will be compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Slope of change in dentate nuclei magnetic susceptibility | Baseline to 24 months
  Magnetic susceptibility of the dentate nuclei will be measured using T2*-weighted multiecho magnetic resonance imaging and quantitative susceptibility mapping processing. The within-person slope of dentate nuclei susceptibility over the three study visits will be estimated and compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Baseline dentate volume | Baseline
  Volume of the dentate nuclei will be measured using T2*-weighted multiecho magnetic resonance imaging and quantitative susceptibility mapping processing. Baseline dentate nuclei volume will be compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Slope of change in dentate volume | Baseline to 24 months
  Volume of the dentate nuclei will be measured using T2*-weighted multiecho magnetic resonance imaging and quantitative susceptibility mapping processing. The within-person slope of dentate nuclei volume over the three study visits will be estimated and compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Baseline total cerebellar volume | Baseline
  Total volume of the cerebellum will be measured using T1- and T2-weighted magnetic resonance imaging. Baseline total cerebellar volume will be compared between the Friedreich ataxia and control groups.
Slope of change in total cerebellar volume | Baseline to 24 months
  Total volume of the cerebellum will be measured using T1- and T2-weighted magnetic resonance imaging. The within-person slope of total cerebellar volume over the three study visits will be estimated and compared between the Friedreich ataxia and control groups.
Baseline superior cerebellar peduncle volume | Baseline
  Volume of the superior cerebellar peduncles will be measured using T1- and T2-weighted magnetic resonance imaging. Baseline superior cerebellar peduncle volume will be compared between the Friedreich ataxia and control groups.
Slope of change in superior cerebellar peduncle volume | Baseline to 24 months
  Volume of the superior cerebellar peduncles will be measured using T1- and T2-weighted magnetic resonance imaging. The within-person slope of superior cerebellar peduncle volume over the three study visits will be estimated and compared between the Friedreich ataxia and control groups.
Baseline superior cerebellar peduncle fractional anisotropy | Baseline
  Fractional anisotropy of the superior cerebellar peduncles will be measured using diffusion tensor magnetic resonance imaging. Baseline superior cerebellar peduncle fractional anisotropy will be compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Slope of change in superior cerebellar peduncle fractional anisotropy | Baseline to 24 months
  Fractional anisotropy of the superior cerebellar peduncles will be measured using diffusion tensor magnetic resonance imaging. The within-person slope of superior cerebellar peduncle fractional anisotropy over the three study visits will be estimated and compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Baseline superior cerebellar peduncle mean diffusivity | Baseline
  Mean diffusivity of the superior cerebellar peduncles will be measured using diffusion tensor magnetic resonance imaging. Baseline superior cerebellar peduncle mean diffusivity will be compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Slope of change in superior cerebellar peduncle mean diffusivity | Baseline to 24 months
  Mean diffusivity of the superior cerebellar peduncles will be measured using diffusion tensor magnetic resonance imaging. The within-person slope of superior cerebellar peduncle mean diffusivity over the three study visits will be estimated and compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Baseline superior cerebellar peduncle radial diffusivity | Baseline
  Radial diffusivity of the superior cerebellar peduncles will be measured using diffusion tensor magnetic resonance imaging. Baseline superior cerebellar peduncle radial diffusivity will be compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Slope of change in superior cerebellar peduncle radial diffusivity | Baseline to 24 months
  Radial diffusivity of the superior cerebellar peduncles will be measured using diffusion tensor magnetic resonance imaging. The within-person slope of superior cerebellar peduncle radial diffusivity over the three study visits will be estimated and compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Baseline superior cerebellar peduncle axial diffusivity | Baseline
  Axial diffusivity of the superior cerebellar peduncles will be measured using diffusion tensor magnetic resonance imaging. Baseline superior cerebellar peduncle axial diffusivity will be compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Slope of change in superior cerebellar peduncle axial diffusivity | Baseline to 24 months
  Axial diffusivity of the superior cerebellar peduncles will be measured using diffusion tensor magnetic resonance imaging. The within-person slope of superior cerebellar peduncle axial diffusivity over the three study visits will be estimated and compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Baseline cervical spinal cord cross-sectional area | Baseline
  Cross-sectional area of the cervical portion of the spinal cord will be measured using T2-weighted magnetic resonance imaging. Baseline cervical spinal cord cross-sectional area will be compared between the Friedreich ataxia and control groups.
Slope of change in cervical spinal cord cross-sectional area | Baseline to 24 months
  Cross-sectional area of the cervical portion of the spinal cord will be measured using T2-weighted magnetic resonance imaging. The within-person slope of cervical spinal cord cross-sectional area over the three study visits will be estimated and compared between the Friedreich ataxia and control groups.
Baseline cervical spinal cord fractional anisotropy | Baseline
  Fractional anisotropy of the cervical portion of the spinal cord will be measured using diffusion tensor magnetic resonance imaging. Baseline cervical spinal cord fractional anisotropy will be compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Slope of change in cervical spinal cord fractional anisotropy | Baseline to 24 months
  Fractional anisotropy of the cervical portion of the spinal cord will be measured using diffusion tensor magnetic resonance imaging. The within-person slope of cervical spinal cord fractional anisotropy over the three study visits will be estimated and compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Baseline cervical spinal cord mean diffusivity | Baseline
  Mean diffusivity of the cervical portion of the spinal cord will be measured using diffusion tensor magnetic resonance imaging. Baseline cervical spinal cord mean diffusivity will be compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Slope of change in cervical spinal cord mean diffusivity | Baseline to 24 months
  Mean diffusivity of the cervical portion of the spinal cord will be measured using diffusion tensor magnetic resonance imaging. The within-person slope of cervical spinal cord mean diffusivity over the three study visits will be estimated and compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Baseline cervical spinal cord radial diffusivity | Baseline
  Radial diffusivity of the cervical portion of the spinal cord will be measured using diffusion tensor magnetic resonance imaging. Baseline cervical spinal cord radial diffusivity will be compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Slope of change in cervical spinal cord radial diffusivity | Baseline to 24 months
  Radial diffusivity of the cervical portion of the spinal cord will be measured using diffusion tensor magnetic resonance imaging. The within-person slope of cervical spinal cord radial diffusivity over the three study visits will be estimated and compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Baseline cervical spinal cord axial diffusivity | Baseline
  Axial diffusivity of the cervical portion of the spinal cord will be measured using diffusion tensor magnetic resonance imaging. Baseline cervical spinal cord axial diffusivity will be compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Slope of change in cervical spinal cord axial diffusivity | Baseline to 24 months
  Axial diffusivity of the cervical portion of the spinal cord will be measured using diffusion tensor magnetic resonance imaging. The within-person slope of cervical spinal cord axial diffusivity over the three study visits will be estimated and compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Baseline cervical spine tNAA/mIns ratio | Baseline
  The ratio of N-acetylaspartate (tNAA) and myo-inositol (mIns) within cervical spinal cord will be measured using sLASER magnetic resonance spectroscopy. The baseline tNAA/mIns ratio will be compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.
Slope of the cervical spine tNAA/mIns ratio | Baseline to 24 months
  The ratio of N-acetylaspartate (tNAA) and myo-inositol (mIns) within cervical spinal cord will be measured using sLASER magnetic resonance spectroscopy. The within-person slope of the tNAA/mIns ratio over the three study visits will be estimated and compared between the Friedreich ataxia and control groups. This measurement will be obtained for participants aged 11 years and over.

SECONDARY OUTCOMES:
Modified Friedreich Ataxia Rating Scale (mFARS) score | Baseline to 24 months
  The modified Friedreich Ataxia Rating Scale (mFARS) is a neurological rating scale comprising four subscales (bulbar, upper limb coordination, lower limb coordination, and upright stability). The total score ranges from 0 to 93, with a higher score reflecting greater neurological severity. This assessment will be administered to participants with FA only.
Upright Stability (US) score | Baseline to 24 months
  The Upright Stability (US) assessment is part of the neurological examination within the Modified Friedreich Ataxia Rating Scale (mFARS). This component comprises nine items: sitting position, stance with feet apart, stance with feet apart and eyes closed, stance with feet together, stance with feet together and eyes closed, tandem stance, stance with dominant foot, tandem walk, and gait. The score ranges from 0 to 9, with a higher score reflecting poorer upright stability (i.e., greater neurological severity). This assessment will be administered to participants with FA only.
Activities of Daily Living (ADL) score | Baseline to 24 months
  Activities of Daily Living (ADL) is a component of the Friedreich Ataxia Rating Scale (FARS), a clinical rating scale developed for FA. The ADL score aims to quantify essential and routine aspects of self-care, often reported on by a family member or caregiver of a person with FA. The ADL comprises 9 items: speech, swallowing, cutting food and handling utensils, dressing, personal hygiene, falling, walking, quality of sitting position, and bladder function. The score ranges from 0 to 36, with a higher score reflecting greater difficulty completing activities of daily living independently. This assessment will be administered to participants with FA only.
Scale for the Assessment and Rating of Ataxia (SARA) score | Baseline to 24 months
  The SARA is a semi-quantitative assessment of ataxia, measuring ataxia of upper limb, lower limb, gait, balance and speech. It has eight items: gait, stance, sitting, speech disturbance, finger chase, nose-finger test, fast alternating hand movement, and heel-shin slide. The total score ranges from 0 (no ataxia) to 40 (severe ataxia). This assessment will be administered to participants with FA only.
9 Hole Peg Test times | Baseline to 24 months
  The 9 Hole Peg Test (9HPT) examines finger dexterity and involves placing and removing nine pegs in a pegboard in the quickest possible time. Two consecutive trials of the dominant hand, followed immediately by two consecutive trials of the non-dominant hand, are undertaken. The average time taken to complete the task, for each of the dominant and non-dominant hand, is calculated. The 9HPT has high intra- and inter-rater reliability and is the most commonly used measure of upper limb function in FA. This assessment will be administered to participants with FA only.
Speech analysis scores | Baseline to 24 months
  A battery of speech evaluations will be administered and recorded on a laptop for analysis, using Redenlab software. This will include: reading of a phonetically-balanced passage, sustained vowel sound, listing days of the week, repeating syllables, and a monologue task. This will form a measure of dysarthria. Redenlab is a US-Australian speech-testing company, https://redenlab.com. This assessment will be administered to participants with FA and controls.
Low-Contrast Sloan Letter Chart (LCSLC) test score | Baseline to 24 months
  Contrast letter acuity for vision will be assessed using back-lit Low-Contrast Sloan Letter Charts (LCSLCs). Participants will sit at an eye distance of 2 metres from the chart. Binocular vision will be assessed using participants' normal corrective lenses where relevant. Participants are required to read each letter on the chart. Three charts will be presented, with three different visual contrast levels: 100% (equivalent to high-contrast visual acuity), 2.5%, and 1.25%. The maximum total score across the three charts (number of letters read correctly) is 240. Scores for each individual chart will also be recorded. This assessment will be administered to participants with FA only.
Cerebellar Cognitive Affective/Schmahmann Syndrome (CCAS) scale score | Baseline to 24 months
  The Cerebellar Cognitive Affective/Schmahmann Syndrome (CCAS) Scale is a 10-item screening measure assessing attention and concentration, executive functioning, memory, language, visuospatial functioning, abstract thinking, and neuropsychiatric features. Each item has an associated raw score and pass/fail evaluation. The total raw score (maximum 120) and the total number of "failed" items (maximum 10) will be recorded. This scale is to be administered to participants who are aged 18 years and over. This assessment will be administered to participants with FA and controls.
Hayling Sentence Completion Test (HSCT) scores | Baseline to 24 months
  The Hayling Sentence Completion Test (HSCT) is an orally-administered test measuring response initiation and response suppression. In the first section, participants are asked to complete a series of incomplete sentences with a sensible word. In the second section, participants are asked to supply an unrelated word to complete each sentence. Scaled scores for total response latency in each section, a scaled score for errors in the second section, and an overall scale score are calculated. This test is to be administered to participants who are aged 18 years and over. This assessment will be administered to participants with FA and controls.
Hospital Anxiety and Depression Scale (HADS) scores | Baseline to 24 months
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item self-assessment scale designed to screen for states of depression and anxiety and measure the severity of these states. It contains a 7-item subscale for each of Anxiety (HADS-A) and Depression (HADS-D). Possible scores for each of the HADS-Anxiety and HADS-Depression scales range from 0 to 21. Higher scores indicate more severe anxiety and depression. This scale is be administered to participants who are aged 18 year and over. This assessment will be administered to participants with FA and controls.
Junior Hayling Sentence Completion Test (Junior HSCT) scores | Baseline to 24 months
  The Junior Hayling Sentence Completion Test (Junior HSCT) is an orally-administered measure of response initiation and response suppression in children. To be administered to participants who are aged at least 8 years but less than 18 years. This assessment will be administered to participants with FA and controls.
Paediatric Cerebellar Cognitive Affective/Schmahmann Syndrome (CCAS) scale score | Baseline to 24 months
  The Paediatric Cerebellar Cognitive Affective/Schmahmann Syndrome (CCAS) scale is an assessment of the executive, visual-spatial and linguistic components of cognitive control and affect in children. Currently under development. To be incorporated as a secondary outcome measure if available at the time of study commencement. To be administered to participants who are aged at least 8 years but less than 18 years. This assessment will be administered to participants with FA and controls.
Revised Children's Anxiety and Depression scale (RCADS) scores | Baseline to 24 months
  The Revised Child Anxiety and Depression Scale (RCADS) is a 47-item, self-report questionnaire six subscales: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and major depressive disorder. It also yields a Total Anxiety Scale and a Total Internalizing Scale. A higher score indicates a higher level of the given disorder/syndrome. This scale is to be administered to participants who are aged at least 8 years but less than 18 years. This assessment will be administered to participants with FA and controls.

OTHER OUTCOMES:
Serum neurofilament light chain (NfL) level | Baseline to 24 months
  Neurofilament light chain (NfL) is a peripherally-accessible blood biomarker of neuroaxonal destruction in various neurodegenerative diseases. It has been shown for several such diseases that blood NfL might serve as a progression biomarker as well as a treatment response biomarker. Blood samples will be collected at each of the three study visits, stored locally, and shipped to a central location for analysis of NfL levels.
Frataxin protein level | Baseline to 24 months
  Levels of frataxin protein in lymphocyte and serum will be measured. Frataxin is produced at reduced levels in FA as a consequence of the guanine-adenine-adenine (GAA) repeat expansion in the frataxin gene (FXN) on chromosome 9. Blood samples will be collected at each of the three study visits, stored locally, and shipped to a central location for analysis of frataxin levels.

CONTACTS AND LOCATIONS:
Overall Officials: Nellie Georgiou-Karistianis, PhD, Principal Investigator — Monash University
Locations (7):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Center for Magnetic Resonance Research, University of Minnesota, Minneapolis, Minnesota
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Monash Biomedical Imaging, Monash University, Clayton, Victoria, Australia
- Lab of Neuroimaging and Dept of Neurology, University of Campinas (UNICAMP), São Paulo, São Paulo, Brazil
- McGill University, Montreal, Quebec, Canada
- Department of Neurology, RWTH Aachen University, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Yes
It is recognised that this project will generate data that is of interest to the FA academic and bio-pharmaceutical, drug development community. All such data (de-identified) will be made available to third parties at the completion of the study after request, with approval from the TRACK-FA Steering Committee. Each site will be required to ensure that participants are consented in such a way that allows the sharing of de-identified data with the community in this manner.
Time Frame: Data will become available after the conclusion of the TRACK-FA study. The study will be 5 years in duration and each academic site may have a slightly different start and end date.
Access Criteria: Data access will be granted on a case-by-case basis after the study has been completed. The requesting party will be required to submit a formal request to the TRACK-FA Steering Committee outlining how the data is to be used and for what purpose.
URL: https://www.monash.edu/medicine/trackfa/news

REFERENCES:
- [Derived] Shiraishi DH, Saha S, Adanyeguh IM, Cocozza S, Corben LA, Deistung A, Delatycki MB, Dogan I, Gaetz W, Georgiou-Karistianis N, Graf S, Grisoli M, Henry PG, Jarola GM, Joers JM, Langkammer C, Lenglet C, Li J, Lobo CC, Lock EF, Lynch DR, Mareci TH, Martinez ARM, Monti S, Nigri A, Pandolfo M, Reetz K, Roberts TP, Romanzetti S, Rudko DA, Scaravilli A, Schulz JB, Subramony SH, Timmann D, Franca MC, Harding IH, Rezende TJR; TRACK-FA Neuroimaging Consortium. Automated Deep Learning-based Segmentation of the Dentate Nucleus Using Quantitative Susceptibility Mapping MRI. Radiol Artif Intell. 2025 Nov;7(6):e240478. doi: 10.1148/ryai.240478. PMID 40767617
- [Derived] Georgiou-Karistianis N, Corben LA, Lock EF, Bujalka H, Adanyeguh I, Corti M, Deelchand DK, Delatycki MB, Dogan I, Farmer J, Franca MC Jr, Gabay AS, Gaetz W, Harding IH, Joers J, Lax MA, Li J, Lynch DR, Mareci TH, Martinez ARM, Pandolfo M, Papoutsi M, Parker RG, Reetz K, Rezende TJR, Roberts TP, Romanzetti S, Rudko DA, Saha S, Schulz JB, Subramony SH, Supramaniam VG, Lenglet C, Henry PG. Neuroimaging Biomarkers for Friedreich Ataxia: A Cross-Sectional Analysis of the TRACK-FA Study. Ann Neurol. 2025 Aug;98(2):386-397. doi: 10.1002/ana.27237. Epub 2025 Mar 22. PMID 40119735
- [Derived] Georgiou-Karistianis N, Corben LA, Reetz K, Adanyeguh IM, Corti M, Deelchand DK, Delatycki MB, Dogan I, Evans R, Farmer J, Franca MC, Gaetz W, Harding IH, Harris KS, Hersch S, Joules R, Joers JJ, Krishnan ML, Lax M, Lock EF, Lynch D, Mareci T, Muthuhetti Gamage S, Pandolfo M, Papoutsi M, Rezende TJR, Roberts TPL, Rosenberg JT, Romanzetti S, Schulz JB, Schilling T, Schwarz AJ, Subramony S, Yao B, Zicha S, Lenglet C, Henry PG. A natural history study to track brain and spinal cord changes in individuals with Friedreich's ataxia: TRACK-FA study protocol. PLoS One. 2022 Nov 21;17(11):e0269649. doi: 10.1371/journal.pone.0269649. eCollection 2022. PMID 36410013
- [Derived] Hernandez ALCC, Rezende TJR, Martinez ARM, de Brito MR, Franca MC Jr. Tract-Specific Spinal Cord Diffusion Tensor Imaging in Friedreich's Ataxia. Mov Disord. 2022 Feb;37(2):354-364. doi: 10.1002/mds.28841. Epub 2021 Oct 29. PMID 34713932